CLINICAL TRIAL: NCT05023889
Title: Spectrum of Peripheral and Autonomic Neuropathies in Patients With aTTRwt Amyloidosis and Response to Patisiran Therapy
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Austin Neuromuscular Center (Other)
Collaborators: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 001 amendment 02
Record Dates: First submitted 2021-08-11; First posted 2021-08-27 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Polyneuropathies; Wild Type ATTR Amyloidosis; Wild-Type Transthyretin-Related (ATTR)Amyloidosis; Wild-Type Transthyretin Cardiac Amyloidosis; Transthyretin Amyloidosis
MeSH Terms: conditions — Polyneuropathies; Amyloid Neuropathies, Familial; Amyloidosis, Hereditary, Transthyretin-Related | interventions — patisiran

STUDY DESIGN:
Intervention Model Description: This protocol is a single center pilot study designed to evaluate the efficacy and safety of patisiran in adult patients with wtATTR amyloidosis and symptomatic polyneuropathy as assessed with Neuropathy Impairment Score (NIS).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- open label (Other): single open arm label
  Interventions: Drug: patisiran

INTERVENTIONS:
Drug: patisiran — Patients will receive 0.3 mg/kg patisiran once every 21 days administered as an IV infusion over 70 minutes (approximately 1 mL/minute for the first 15 minutes followed by approximately 3 mL/minute for the remainder of the infusion) by a controlled infusion device.
  All patients in this study will be premedicated prior to dosing with patisiran. Study drug supplied for this study must not be used for any purpose other than the present study and must not be administered to any person not enrolled in the study.
  The first dose of study drug (week 1) will be administered under the supervision of site personnel. After the first dose of patisiran, patients should return to the site for patisiran dosing once every 21 days or receive the patisiran infusions at a local infusion center by a healthcare professional trained on the Protocol, administration of premedication, and patisiran infusion. Patient must receive a dose of interventional drug within the dosing window (±3 days).
  Other Names: ONPATTRO

SUMMARY:
To evaluate the efficacy and safety of patisiran in patients with wtATTR amyloidosis and symptomatic polyneuropathy by evaluating the effect on neurologic impairment and quality of life.

DETAILED DESCRIPTION:
The study will consist of a baseline screening period and a 24-month treatment period. Eligible patient will receive patisiran administered as an IV infusion once every 21 days for a 24-month period. During the 24-month treatment period study patients will undergo assessments for efficacy and/or safety as outlined in the schedule of assessments with key efficacy assessments being performed prior to the first dose and proceeding as outlined in the schedule of assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female >18
2. Diagnosis of symptomatic polyneuropathy
3. wtATTR based on cardiac biopsy or Tc99m PYP
4. Negative hATTR sequencing
5. 0 to 0.5 gram/dl serum monoclonal protein.
6. No history of other secondary causes of neuropathy.
7. Have adequate complete blood counts and liver function tests
8. Have negative serology for hepatitis B virus (HBV) and hepatitis C virus (HCV)

Exclusion Criteria:

1. Other Causes of neuropathy as determined by the principle investigator.
2. Has known human immunodeficiency virus (HIV) infection;
3. Primary AL.
4. NYHA Class IV at the Screening visit. 5. Has any of the following laboratory parameter assessments at screening:

   1. Aspartate transaminase (AST) or alanine transaminase (ALT) levels ˃2.0 × the upper limit of normal (ULN).
   2. Total bilirubin ˃ULN. Patients with elevated total bilirubin that is secondary to documented Gilbert's syndrome are eligible if total bilirubin <2 × ULN.
   3. International normalized ratio (INR) ˃1.5 (unless patient is on anticoagulant therapy, in which case excluded if INR ˃3.5).

      6. Has eGFR < 30 mL/min/1.73 m2 (using the modification of diet in renal disease [MDRD] formula). 7. Is currently taking diflunisal; if previously on this agent, must have at least a 6-month wash-out prior to dosing (Day 1).

      8. Is currently taking doxycycline, or tauroursodeoxycholic acid; if previously on any of these agents must have completed a 30-day wash-out prior to dosing (Day 1).

      9. Received prior TTR-lowering treatment or participated in a gene therapy trial for amyloidosis. 10. Current or future participation in another investigational device or drug study, Scheduled to occur during this study, or has received an investigational agent or device within 30 days (or 5 half-lives of the investigational drug, whichever is longer) prior to dosing (Day 1). In the case of investigational TTR stabilizer drugs, washout for 6 months prior to dosing (Day 1) is required; this does not apply to patients who are on tafamidis at baseline (per inclusion Criterion 4).

      11. Requires treatment with calcium channel blockers (eg, verapamil, diltiazem) or digitalis.

      12. Other non-TTR cardiomyopathy, hypertensive cardiomyopathy, cardiomyopathy due to valvular heart disease, or cardiomyopathy due to ischemic heart disease.

      13. Has non-amyloid disease affecting exercise testing (eg, severe chronic obstructive pulmonary disease, severe arthritis, or peripheral vascular disease affecting ambulation).

      14. Had acute coronary syndrome or unstable angina within the past 3 months. 15. Has history of sustained ventricular tachycardia or aborted ventricular fibrillation.

      16. Has persistent elevation of systolic (˃180 mmHg) and diastolic (˃100 mmHg) blood pressure that is considered uncontrolled by physician.

17-Has untreated hypo- or hyperthyroidism. 18-Prior or planned heart, liver, or other organ transplant. 19. Had a malignancy within 5 years, except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated.

20. Has other medical conditions or comorbidities which, in the opinion of the Investigator would interfere with study compliance or data interpretation. 21. Female Is not willing to comply with the contraceptive requirements during the study period.

22. History of illicit drug abuse within the past 5 years that in the opinion of the Investigator would interfere with compliance with study procedures or follow-up visits.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2026-02-19 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
Change in Neurological Impairment Score | baseline to 24 months
  to assess the severity of functional impairment of motor and sensory nerves.NIS is a measure of motor strength, comprised of cranial nerve and both upper and lower limb motor assessments. The minimum and maximum values are 0 and 192, respectively. A higher score indicates a worse outcome.
Norfolk QOL-DN | baseline to 24 months
  Change in Norfolk Quality of Life Questionnaire (Norfolk QOL-DN).The change from baseline in Norfolk QoL-DN at 24 months. The Norfolk QoL-DN questionnaire is a standardized 35-item patient-reported outcomes measure of diabetic neuropathy - small fiber, large fiber, and autonomic nerve function. The minimum and maximum values are -4 and 136, respectively. A higher score indicates a worse outcome.
COMPASS 31score | baseline to 24 months
  Composite Autonomic Symptom Score (COMPASS) 31a self-assessment instrument for patient reported autonomic symptoms such as dizziness, constipation, diarrhea, nausea/vomiting, and incontinence. The minimum and maximum values are 0 and 100, respectively. A higher score indicates a worse outcome

SECONDARY OUTCOMES:
PND Polyneuropathy disability (PND) Score | baseline to 24 months
  To compare and identify changes. Stage 0: no impairment Stage I: sensory disturbances but preserved walking capability Stage II: impaired walking capability but ability to walk without a stick or crutches Stage III a: walking only with the help of one stick or crutch Stage III b: walking with the help of two sticks or crutches. V: confined to wheelchair or bedridden A higher score indicates a worse outcome.
Karnofsky, performance status score | baseline to 24 months
  Karnofsky performance score is 11 level score which ranges between 0 (death) to 100 (no evidence of disease). Higher score means higher ability to perform daily tasks.
EuroQOL | baseline to 24 months
  EuroQOL,- A measurement tool that assesses generic quality of life in mobility, self-care, usual activities, pain/discomfort, anxiety/depression The minimum and maximum values are 0 and 100, respectively. A higher score indicates a worse outcome.
EMG -Electromyography | baseline to 24 months
  (EMG) is a diagnostic test that measures how the muscles and nerves work to evaluate peripheral Neuropathies pattern and progression
Tilt Table Test | 24 months
  Evaluate and compare the response of blood pressure and heart rate changes in posture and position.
Optional exploratory nerve and muscle biopsy | during screening visit ( 28 day window)
  to identify amyloid deposits in skeletal muscle and peripheral nerve

OTHER OUTCOMES:
Cardiac MRI | start of study, and study end at 2 years
  to identify cardiac abnormalities or changes and comparison
Echo with strain | start of study, and study end at 2 years
  to identify cardiac abnormalities or changes and comparison
PYP - mTc99-PYP | start of study, and study end at 2 years
  for cardiac amyloidosis imaging. - to identify cardiac function changes and comparison
NT Pro BNP blood draw | start of study, and study end at 2 years
  serum biomarker to evaluate heart failure severity, ( pg/ml)
NFL blood draw | at start, month 1,2,3,6 and every 6 months after until study end at two years
  Serum Neurofilament Light Chain level in patients with evolving disease, ( pg/mL)

CONTACTS AND LOCATIONS:
Locations (1):
- Austin Neuromuscler Center/National Neuromuscular Research Institute, Austin, Texas, United States